CLINICAL TRIAL: NCT06352502
Title: Efficacy and Safety of Furmonertinib for Epidermal Growth Factor Receptor (EGFR) Sensitive Mutation Positive Non-Small Cell Lung Cancer (NSCLC) Patients With Brain Metastasis: a Prospective Observational Study
Brief Title: An Observational Study of Furmonertinib for EGFR Mutation-positive NSCLC Patients With Brain Metastasis
Status: Recruiting | Type: Observational
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 202112-28
Record Dates: First submitted 2024-03-07; First posted 2024-04-08 (Actual); Last update posted 2024-04-08 (Actual); Status verified 2024-04

CONDITIONS: EGF-R Positive Non-Small Cell Lung Cancer; CNS Metastases
Keywords: EGFR; NSCLC; Furmonertinib; CNS metastases
MeSH Terms: interventions — aflutinib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Furmonertinib group: Patients treated with Furmonertinib
  Interventions: Drug: Furmonertinib

INTERVENTIONS:
Drug: Furmonertinib — Patients treated with Furmonertinib mesilate tablets orally
  Other Names: AST2818

SUMMARY:
EGFR mutation positive advanced NSCLC patients with CNS metastases were associated with poor prognosis. Furmonertinib showed promising CNS efficacy in doses of 80 mg orally once daily or higher in patients with EGFR T790M mutation positive NSCLC. This study aims to investigate the efficacy and safety of furmonertinib in the treatment of EGFR-sensitive mutation positive NSCLC patients with brain metastasis.

DETAILED DESCRIPTION:
This study aims to prospectively observe the efficacy and safety of furmonertinib in the treatment of EGFR-sensitive mutation positive NSCLC patients with brain metastasis and will recruit about 30 patients in China.

Furmonertinib (AST2818) is a brain penetrant third generation EGFR TKI. In preclinical studies, the concentration of furmonertinib and its main active metabolite in the brain was higher than that in the plasma, indicating that furmonertinib had the potential to treat CNS metastases. Furmonertinib showed promising CNS efficacy in doses of 80 mg orally once daily in patients with EGFR T790M mutated NSCLC, the median CNS PFS was 11.6 months and 19.3 months in the 80 mg and 160 mg orally once daily group, and the CNS ORR was 65% and 85% in the 80 mg and 160 mg group.

This study will enroll the EGFR-sensitive mutation positive NSCLC patients with brain metastasis who are treated by furmonertinib, and the efficacy and safety data will be recorded.

ELIGIBILITY:
Inclusion Criteria:

1. at least 18 years of age;
2. Histologically or cytologically confirmed metastatic non-squamous Non-Small Cell Lung Cancer (NSCLC);
3. Patient with EGFR 19Del or L858R mutation diagnosed histologically or cytologically.( EGFR L858R or Del 19 with/without T790M )
4. Imaging (MR/CT) confirmed untreated brain metastases before Furmonertinib initiation;
5. Organ function is compatible with oral Furmonertinib therapy (investigator determination based on real-world practice);
6. Life expectancy ≥12 weeks before Fumonertinib initiation;
7. ECOG PS of 0 to 2;
8. Sign the informed consent form.

Exclusion Criteria:

1. Any Third-Epidermal growth factor receptor tyrosine kinase inhibitors (EGFR-TKI) before Furmonertinib initiation;
2. Known hypersensitivity to Furmonertinib or its excipient components;
3. Simultaneous systemic chemotherapy or WBI;
4. The time from the treatment with any other investigational product or its analogue before Furmonertinib initiation does not exceed 5 half-lives of the drug or 14 days, whichever is longer;
5. Any evidence of severe or uncontrolled systemic diseases;
6. Presence of any disease that may strongly interfere with oral drug absorption; presence of any factor that contributes to QTc prolongation or increased risk of arrhythmia; presence of interstitial pneumonitis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with EGFR 19Del or L858R mutation diagnosed histologically or cytologically and imaging (MR/CT) confirmed untreated brain metastases before Furmonertinib initiation.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Estimated)
Dates: Start 2022-01-28 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-09-30 (Estimated)

PRIMARY OUTCOMES:
Intracranial Objective response rate | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 2 years.
  Per Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) using Investigator assessments, is defined as the number (%) of patients with CNS lesion response of Complete Response or Partial Response, will be assessed up to 2 years.
Intracranial Disease Control Rate | Data obtained up until progression, or the last evaluable assessment in the absence of progression, will be assessed up to 2 years.
  The percentage of subjects who have a best CNS lesion response of Complete Response (CR) or Partial Response (PR) or Stable Disease (SD) by Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST 1.1) as assessed by the Investigator, will be assessed up to 2 years.
Intracranial progression-free survival | Intracranial progression-free survival (PFS) analysis based on investigator assessment and will be assessed up to 3 years.
  Intracranial progression-free survival (PFS) analysis based on investigator assessment and will be assessed up to 3 years.

SECONDARY OUTCOMES:
Progression-free survival | Progression-free survival (PFS) analysis based on investigator assessment per RECIST 1.1, and will be assessed up to 2 years.
  Progression-free survival (PFS) is defined as the time from first dose of Furmonertinib recorded until the date of disease progression based on investigator assessment.
Overall Survival | The time from beginning of furmonertinib treatment until death due to any cause and will be assessed up to 3 years.
  Overall survival is defined as the time from beginning of furmonertinib treatment until death due to any cause and will be assessed up to 3 years.
Safety/Adverse event | From the recorded first dose of Furmonertinib to 4 weeks after the recorded last dose of Furmonertinib
  Incidence of Adverse Events (AEs): Incidence, severity and seriousness of adverse events, incidence of serious adverse events (SAEs), which usually be graded by CTCAE v5.0 based on current clinical practice.

CONTACTS AND LOCATIONS:
Overall Officials: Haichuan Su, PhD, Principal Investigator — Tang-Du Hospital
Locations (1):
- Tangdu Hopspital, Xi’an, Shanxi, China

IPD SHARING:
Plan to Share IPD: No